CLINICAL TRIAL: NCT05979337
Title: Brief Behavioral Interventions for Adults With Chronic Migraine
Brief Title: Brief Interventions in Chronic Migraine
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, John Sturgeon, Assistant Professor of Anesthesiology, University of Michigan
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: HUM00237000; 7K23NS125004-02 (NIH)
Record Dates: First submitted 2023-07-28; First posted 2023-08-07 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Chronic Migraine
Keywords: Health Education; Migraine-related disability; Empowered Relief
MeSH Terms: conditions — Health Education | interventions — Therapeutics

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Empowered Relief (ER) class (Experimental): Daily Diaries
  Interventions: Behavioral: Empowered Relief
- Health Education (HE) class (Experimental)
  Interventions: Behavioral: Health Education (HE)
- Empowered Relief (ER) class and Health Education (HE) class (Experimental): If randomized to both classes, the HE class will occur first with a week break in between to the ER class.
  Interventions: Behavioral: Empowered Relief; Behavioral: Health Education (HE)
- Treatment as Usual (TAU) (Other)
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: Empowered Relief — This is a single-session (2-hour) behavioral intervention utilizing pain psychology principles (cognitive-behavioral therapy for pain, pain neuroscience education).
  Class will take place over zoom and have up to 25 participants. The Zoom classes will not be recorded. Participant will be asked to have the camera on during the entire class for treatment course/class validity. Participants are not required to speak during the class but are welcome to ask questions.
  Participants will complete daily diaries for 14 days prior to attending study classes, and another 14 days after completing study classes.
  In addition, participants will complete questionnaires and information about medical and personal history, symptoms, mood, sleep, medication use, and ability to function in daily life.
  Arms: Empowered Relief (ER) class; Empowered Relief (ER) class and Health Education (HE) class
Behavioral: Health Education (HE) — This is a single-session (2-hour) health education class reviewing principles of medically indicated self-management of migraine headaches (e.g., consistent dietary and hydration habits, exercise, understanding of and adherence to medical treatment regimens).
  Class will take place over zoom and have up to 25 participants. The Zoom classes will not be recorded. Participant will be asked to have the camera on during the entire class for treatment course/class validity. Participants are not required to speak during the class but are welcome to ask questions.
  Participants will complete daily diaries for 14 days prior to attending study classes, and another 14 days after completing study classes.
  In addition, participants will complete questionnaires and information about medical and personal history, symptoms, mood, sleep, medication use, and ability to function in daily life.
  Arms: Empowered Relief (ER) class and Health Education (HE) class; Health Education (HE) class
Behavioral: Treatment as Usual — Participants will complete questionnaires and information about medical and personal history, symptoms, mood, sleep, medication use, and ability to function in daily life. In addition, participants will complete daily diaries for 28 days.
  If participants are interested in attending classes that were not part of this group assignment, participants will be invited to do so after completing the 6-month follow-up questionnaire.
  Arms: Treatment as Usual (TAU)

SUMMARY:
People with chronic migraine headaches face many challenges, including high levels of daily pain, disturbances to everyday activities and sleep, and problems with mood such as depression or anxiety. This trial is being completed to study whether changing an individual's behaviors may have an impact as a treatment for migraine headaches.

Eligible participants will be randomized to one of the four arms. This study will be conducted remotely without in-person contact.

Study Hypothesis:

* There is a main effect of attending either the Empowered Relief and Health Education intervention on reductions in migraine-related disability 1 month after completing either intervention
* There is a main effect of Empowered Relief and Health Education interventions on reducing pain-related catastrophizing and migraine symptom severity 1 month after completing either intervention (secondary hypothesis)
* The expected reductions in migraine-related disability, pain catastrophizing, and migraine symptom severity will be maintained at secondary time points (2 months, 3 months, and 6 months after completing either intervention) (secondary hypothesis)

ELIGIBILITY:
Inclusion Criteria:

* Self-reported neurologist diagnosis of chronic migraine
* Meets diagnostic criteria for chronic migraine according to the Identify Chronic Migraine (IDCM) self-reported instrument
* English-speaking
* Internet access and audio-visual conferencing capability (e.g., Zoom meetings by phone or computer) in the home
* Age 18 years or older

Exclusion Criteria:

* Currently receiving cognitive-behavioral therapy for pain or migraine
* Open litigation regarding a medical condition, as assessed in preliminary study screening
* Inability to provide informed consent and complete study procedures (e.g., indications of suspected major cognitive impairment via observations of study staff during consenting) that would preclude comprehension or participation in study protocols
* Failure to complete at least 7 out of 14 pre-intervention daily diaries

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-10-11 (Actual); Primary Completion 2026-04-02 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Change in Migraine Disability Assessment Test - 28 Day Version (MIDAS-28) Scores | Baseline, 1 month
  The MIDAS is a 5-item questionnaire to measure the impact of headaches on life. Subjects indicate how many days headaches have impacted a specific activity. Score ranges: 0-5: little or no disability; 6-10: mild disability; 11-20: moderate disability: 21 (+) severe disability.

SECONDARY OUTCOMES:
Change in Migraine Disability Assessment Test - 28 Day Version (MIDAS-28) Scores | Baseline, 2 months
  The MIDAS-28 is a 5-item questionnaire to measure the impact of headaches on life. Subjects indicate how many days headaches have impacted a specific activity. Score ranges: 0-5: little or no disability; 6-10: mild disability; 11-20: moderate disability: 21 (+) severe disability.
Change in Migraine Disability Assessment Test - 28 Day Version (MIDAS-28) Scores | Baseline, 3 months
  The MIDAS-28 is a 5-item questionnaire to measure the impact of headaches on life. Subjects indicate how many days headaches have impacted a specific activity. Score ranges: 0-5: little or no disability; 6-10: mild disability; 11-20: moderate disability: 21 (+) severe disability.
Change in Migraine Disability Assessment Test - 28 Day Version (MIDAS-28) Scores | Baseline, 6 months
  The MIDAS-28 is a 5-item questionnaire to measure the impact of headaches on life. Subjects indicate how many days headaches have impacted a specific activity. Score ranges: 0-5: little or no disability; 6-10: mild disability; 11-20: moderate disability: 21 (+) severe disability.
Change Migraine Symptom Severity Scale (MSSS) | Baseline, 1 month
  A composite score of 7 self-report questions that incorporates information about headache criteria (unilateral pain, pulsatile pain, moderate, or severe pain intensity, routine activities worsen pain, nausea, photophobia, and phonophobia). The overall MSSS score ranges from 0 to 21 calculated by adding scores ranging from 0 to 3 for each of the 7 headache features assessed.
Change Migraine Symptom Severity Scale (MSSS) | Baseline, 2 month
  A composite score of 7 self-report questions that incorporates information about headache criteria (unilateral pain, pulsatile pain, moderate, or severe pain intensity, routine activities worsen pain, nausea, photophobia, and phonophobia). The overall MSSS score ranges from 0 to 21 calculated by adding scores ranging from 0 to 3 for each of the 7 headache features assessed.
Change Migraine Symptom Severity Scale (MSSS) | Baseline, 3 month
  A composite score of 7 self-report questions that incorporates information about headache criteria (unilateral pain, pulsatile pain, moderate, or severe pain intensity, routine activities worsen pain, nausea, photophobia, and phonophobia). The overall MSSS score ranges from 0 to 21 calculated by adding scores ranging from 0 to 3 for each of the 7 headache features assessed.
Change Migraine Symptom Severity Scale (MSSS) | Baseline, 6 month
  A composite score of 7 self-report questions that incorporates information about headache criteria (unilateral pain, pulsatile pain, moderate, or severe pain intensity, routine activities worsen pain, nausea, photophobia, and phonophobia). The overall MSSS score ranges from 0 to 21 calculated by adding scores ranging from 0 to 3 for each of the 7 headache features assessed.
Change in Pain Catastrophizing Scale (PCS) | Baseline, 1 month
  The PCS has 13 items rated on 5 point scales from 0 (not at all) to 4 (all the time). Total scores range from 0-52. Higher scores are worse.
Change in Pain Catastrophizing Scale (PCS) | Baseline, 2 month
  The PCS has 13 items rated on 5 point scales from 0 (not at all) to 4 (all the time). Total scores range from 0-52. Higher scores are worse.
Change in Pain Catastrophizing Scale (PCS) | Baseline, 3 month
  The PCS has 13 items rated on 5 point scales from 0 (not at all) to 4 (all the time). Total scores range from 0-52. Higher scores are worse.
Change in Pain Catastrophizing Scale (PCS) | Baseline, 6 month
  The PCS has 13 items rated on 5 point scales from 0 (not at all) to 4 (all the time). Total scores range from 0-52. Higher scores are worse.

CONTACTS AND LOCATIONS:
Overall Officials: John Sturgeon, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified datasets including participant self-report data (baseline, follow-up and daily diary-based assessments) will be maintained and made available to external researchers upon request via the Inter-University Consortium for Political and Social Research (ICPSR) data repository at University of Michigan.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: De-identified datasets will be made available after publication of the primary study results and/or at the conclusion of the National Institute of Neurological Disorders and Stroke (NINDS)-funded grant study period (currently December 2026, barring any no-cost extension. Data will remain available for at least 3 years beyond the end date of the study.
Access Criteria: Data may be shared with other investigators interested in learning more about the nature of behavioral interventions for individuals with chronic migraine. All datasets will be de-identified and shared only after interested researchers contact ICPSR and complete a restricted data use agreement.
  The data and associated documentation will be made available to users only under a restricted data-sharing agreement through ICPSR that provides for (a) a commitment to using the data only for research purposes and not to identify any individual participant; (b) a commitment to securing the data using appropriate computer technology; and (c) a commitment to destroying or returning the data after analyses are completed. Such a data-use agreement will be executed through the PI and ICPSR through the University of Michigan.